CLINICAL TRIAL: NCT04820023
Title: A Phase 1/2, Open-Label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of BBT-176 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) Who Progressed Following Prior Therapy With an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR TKI) Agent
Brief Title: Phase 1/2 Study of BBT-176 in Advanced NSCLC With Progression After EGFR TKI Treatment
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision considering the changing treatment landscape for NSCLC
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBT176-ONC-001
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: NSCLC
MeSH Terms: interventions — BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- 20mg QD (Experimental): BBT-176: 20mg, Orally, Once daily (QD)
  Interventions: Drug: BBT-176, QD
- 80mg QD (Experimental): BBT-176: 80mg, Orally, QD
  Interventions: Drug: BBT-176, QD
- 160mg QD (Experimental): BBT-176: 160mg, Orally, QD
  Interventions: Drug: BBT-176, QD
- 320mg QD (Experimental): BBT-176: 320mg, Orally, QD
  Interventions: Drug: BBT-176, QD
- 480mg QD (Experimental): BBT-176: 480mg, Orally, QD
  Interventions: Drug: BBT-176, QD
- 600mg QD (Experimental): BBT-176: 600mg, Orally, QD
  Interventions: Drug: BBT-176, QD
- 160mg, BID (Experimental): BBT-176: 160mg, Orally, Twice daily (BID)
  Interventions: Drug: BBT-176, BID
- 200mg, BID (Experimental): BBT-176: 200mg, Orally, BID
  Interventions: Drug: BBT-176, BID
- 240mg, BID (Experimental): BBT-176: 240mg, Orally, BID
  Interventions: Drug: BBT-176, BID

INTERVENTIONS:
Drug: BBT-176, QD — BBT-176 given orally alone, QD
  Arms: 160mg QD; 20mg QD; 320mg QD; 480mg QD; 600mg QD; 80mg QD
Drug: BBT-176, BID — BBT-176 given orally alone, BID
  Arms: 160mg, BID; 200mg, BID; 240mg, BID

SUMMARY:
This clinical trial is the first-in-human study of BBT-176. The purpose of this trial is to investigate the safety and tolerability of BBT-176 (Part 1) and to evaluate the anti-tumor activity of BBT-176 (Part 2).

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of signed and dated, written informed consent before any study specific procedures, sampling and analyses
* Histological or cytological confirmation of advanced and/or metastatic stage IIIB/IV NSCLC
* Radiological documentation of disease progression while on a previous continuous (at least 30 days) treatment with an EGFR TKI monotherapy (including, but not limited to, osimertinib, afatinib, gefitinib, or erlotinib)
* Patients must fulfill one of the following:

  * Confirmation that the tumor harbors an EGFR mutation known to be associated with EGFR TKI sensitivity (including, but not limited to, exon 19 deletion, L858R, or L861Q)
  * Documented partial or complete response or a significant and durable stable disease (at least 6 months), based on the RECIST or WHO criteria, after treatment of an EGFR TKI

Key Exclusion Criteria:

* Treatment with any of the following:

  * An EGFR TKI, including but not limited to osimertinib, afatinib, gefitinib, or erlotinib within 8 days of the first dose of study treatment.
  * Any cytotoxic chemotherapy, investigational agents, or anticancer drugs for the treatment of advanced NSCLC, between prior EGFR TKI treatment and BBT-176 treatment
  * Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
  * Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment
  * Patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation within 6 weeks of the first dose of study treatment
* Any unresolved toxicities from prior therapy greater than NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0) Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2 neuropathy related to prior platinum-therapy
* Spinal cord compression or brain metastases, unless asymptomatic and stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

REFERENCES:
- [Derived] Lim SM, Fujino T, Kim C, Lee G, Lee YH, Kim DW, Ahn JS, Mitsudomi T, Jin T, Lee SY. BBT-176, a Novel Fourth-Generation Tyrosine Kinase Inhibitor for Osimertinib-Resistant EGFR Mutations in Non-Small Cell Lung Cancer. Clin Cancer Res. 2023 Aug 15;29(16):3004-3016. doi: 10.1158/1078-0432.CCR-22-3901. PMID 37249619

RESULTS

PARTICIPANT FLOW:
Groups:
- 20mg QD: BBT-176: 20mg, Orally, QD
- 160mg, QD: BBT-176: 160mg, Orally, QD
- 320mg, QD: BBT-176: 320mg, Orally, QD
- 480mg, QD: BBT-176: 480mg, Orally, QD
- 600mg, QD: BBT-176: 600mg, Orally, QD
- 160mg, BID: BBT-176: 160mg, Orally, BID
Period: Overall Study
Arm/Group | 20mg QD | 80mg QD | 160mg, QD | 320mg, QD | 480mg, QD | 600mg, QD | 160mg, BID | 200mg, BID | 240mg, BID
Started | 4 | 3 | 4 | 3 | 8 | 3 | 5 | 9 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 4 | 3 | 8 | 3 | 5 | 9 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 1 | 4 | 3 | 3 | 6 | 5
Not completed — Progressive Disease | 3 | 0 | 2 | 2 | 2 | 0 | 1 | 1 | 0
Not completed — New anti-cancer therapy | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Each treatment cycle is 21 days.
Groups:
- 160mg BID: BBT-176: 160mg, Orally, BID
- 200mg BID: BBT-176: 200mg, Orally, BID
- 240mg BID: BBT-176: 240mg, Orally, BID
- Total: Total of all reporting groups
Arm/Group | 20mg QD | 80mg QD | 160mg QD | 320mg QD | 480mg QD | 600mg QD | 160mg BID | 200mg BID | 240mg BID | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 8 | 3 | 5 | 9 | 6 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (6.5) | 62.3 (11.9) | 48.0 (9.1) | 50.0 (10.1) | 63.9 (10.1) | 73.0 (5.3) | 63.2 (9.4) | 62.3 (10.5) | 65.5 (7.1) | 62.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 2 | 6 | 2 | 2 | 7 | 5 | 31
  Male | 1 | 0 | 3 | 1 | 2 | 1 | 3 | 2 | 1 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 4 | 3 | 8 | 3 | 5 | 9 | 6 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: (Part 1) Incidence of Adverse Events and Clinical Laboratory Abnormalities Defined as Dose-limiting Toxicities (DLTs)
Description: Any toxicity not attributable to the disease or disease-related processes under investigation that occurs from the first dose of study treatment in dose-escalation cohorts as defined in the protocol.
Time Frame: 21 days from the first dosing
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg QD | 80mg QD | 160mg, QD | 320mg, QD | 480mg, QD | 600mg, QD | 160mg, BID | 200mg, BID | 240mg, BID
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 8 | 3 | 5 | 9 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

2. Primary Outcome: (Part 2) Objective Response Rate (ORR)
Description: ORR is estimated by the number of patients with a best overall response of CR or PR divided by the total number of patients who are evaluable for efficacy.
Time Frame: Every 6 weeks
Population: Due to early termination of the study, Part 2 and analysis was not conducted.
Groups:
- BBT-176: BBT-176: BBT-176 given orally alone
Arm/Group | BBT-176
Number analyzed (Participants) | 0

3. Secondary Outcome: (Part 1) Objective Response Rate (ORR)
Description: ORR is estimated by the number of patients with a best overall response of Complete Response (CR) or Partial Response (PR) divided by the total number of patients who are evaluable for efficacy.
Time Frame: Every 6 weeks, approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 20mg QD | 80mg QD | 160mg, QD | 320mg, QD | 480mg, QD | 600mg, QD | 160mg, BID | 200mg, BID | 240mg, BID
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 8 | 3 | 5 | 9 | 6
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: (Part 1) Pharmacokinetics (PK) Parameters - Peak Concentration (Cmax)
Description: Peak plasma concentration (Cmax) of BBT-176 from Part 1.
Time Frame: 0, 1, 2, 4, 6, 8, 12 hours post-dose on Cycle 1 Day 1 (C1D1) and Cycle 2 Day 1 (C2D1) (each cycle is 21 days)
Population: The presentation of PK data on C1D1 and C2D1 was due to that the PK samples were collected on those dates.
  PK samples were collected at 600 mg QD, but drug exposure was low due to vomiting, making it impossible to determine PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 20mg QD C1D1: BBT-176: 20mg QD C1D1
- 20mg QD C2D1: BBT-176: 20mg QD C2D1
- 80mg QD C1D1: BBT-176: 80mg QD C1D1
- 80mg QD C2D1: BBT-176: 80mg QD C2D1
- 160mg QD C1D1: BBT-176: 160mg QD C1D1
- 160mg QD C2D1: BBT-176: 160mg QD C2D1
- 320mg QD C1D1: BBT-176: 320mg QD C1D1
- 320mg QD C2D1: BBT-176: 320mg QD C2D1
- 480mg QD C1D1: BBT-176: 480mg QD C1D1
- 480mg QD C2D1: BBT-176: 480mg QD C2D1
- 600mg QD C1D1: BBT-176: 600mg QD C1D1
  - PK samples were collected at 600 mg QD, but drug exposure was low due to vomiting, making it impossible to determine PK parameters.
- 600mg QD C2D1: BBT-176: 600mg QD C2D1
  - PK samples were collected at 600 mg QD, but drug exposure was low due to vomiting, making it impossible to determine PK parameters.
- 160mg BID C1D1: BBT-176: 160mg BID C1D1
- 160mg BID C2D1: BBT-176: 160mg BID C2D1
- 200mg BID C1D1: BBT-176: 200mg BID C1D1
- 200mg BID C2D1: BBT-176: 200mg BID C2D1
- 240mg BID C1D1: BBT-176: 240mg BID C1D1
- 240mg BID C2D1: BBT-176: 240mg BID C2D1
Arm/Group | 20mg QD C1D1 | 20mg QD C2D1 | 80mg QD C1D1 | 80mg QD C2D1 | 160mg QD C1D1 | 160mg QD C2D1 | 320mg QD C1D1 | 320mg QD C2D1 | 480mg QD C1D1 | 480mg QD C2D1 | 600mg QD C1D1 | 600mg QD C2D1 | 160mg BID C1D1 | 160mg BID C2D1 | 200mg BID C1D1 | 200mg BID C2D1 | 240mg BID C1D1 | 240mg BID C2D1
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 3 | 3 | 8 | 3 | 3 | 2 | 5 | 3 | 8 | 4 | 6 | 3
ng/mL | 7 (4) | 10 (5) | 159 (67) | 260 (37) | 240 (75) | 638 (231) | 594 (94) | 1416 (370) | 1087 (470) | 2145 (1438) | NA (NA) — c. PK samples were collected at 600 mg QD, but values were low or below the level of detection due to vomiting. The sample numbers with measured concentrations were insufficient to determine the PK parameters. | NA (NA) — c. PK samples were collected at 600 mg QD, but values were low or below the level of detection due to vomiting. The sample numbers with measured concentrations were insufficient to determine the PK parameters. | 255 (80) | 1186 (695) | 354 (88) | 1784 (358) | 399 (154) | 1622 (472)

5. Secondary Outcome: (Part 1) PK Parameters - Area Under the Concentration-time Curve (AUC)
Description: Area under the plasma concentration-time curve (AUC) of BBT-176 from Part 1.
Time Frame: 0, 1, 2, 4, 6, 8, 12 hours post-dose on Cycle 1 Day 1 (C1D1) and Cycle 2 Day 1 (C2D1) (each cycle is 21 days)
Population: PK data were presented on C1D1 and C2D1 as samples were collected on those days. In the BID regimen, AUC 0-12 was calculated on both days. AUC 0-24 was estimated on C2D1 using AUC 0-12, assuming steady state, but not on C1D1 since steady state was not reached. In Cohort 6 (600mg QD), PK parameters were not determined as BBT-176 was not tolerable, and drug exposure was low due to vomiting.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- 600mg QD C1D1: BBT-176: 600mg QD C1D1
- 600mg QD C2D1: BBT-176: 600mg QD C2D1
Arm/Group | 20mg QD C1D1 | 20mg QD C2D1 | 80mg QD C1D1 | 80mg QD C2D1 | 160mg QD C1D1 | 160mg QD C2D1 | 320mg QD C1D1 | 320mg QD C2D1 | 480mg QD C1D1 | 480mg QD C2D1 | 600mg QD C1D1 | 600mg QD C2D1 | 160mg BID C2D1 | 200mg BID C2D1 | 240mg BID C2D1
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 3 | 3 | 8 | 3 | 3 | 2 | 3 | 4 | 3
ng*hr/mL | 91 (42) | 192 (89) | 1314 (263) | 3584 (158) | 2799 (1030) | 9652 (5978) | 8065 (2703) | 21992 (5494) | 13938 (6315) | 38365 (21815) | NA (NA) — c. PK samples were collected at 600 mg QD, but values were low or below the level of detection due to vomiting. The sample numbers with measured concentrations were insufficient to determine the PK parameters. | NA (NA) — c. PK samples were collected at 600 mg QD, but values were low or below the level of detection due to vomiting. The sample numbers with measured concentrations were insufficient to determine the PK parameters. | 20842 (11511) | 37564 (8612) | 33521 (9070)

6. Secondary Outcome: (Part 2) Duration of Response (DoR)
Description: DoR is calculated for every patient with a response to therapy (PR and CR) and is defined as the number of days from the date of initial response to the date of the first documented disease progression/relapse (including clinical progression) or death, whichever occurs first.
Time Frame: throughout study completion, approximately 1 year
Population: Due to early termination of the study, Part 2 and analysis was not conducted.
Arm/Group | BBT-176
Number analyzed (Participants) | 0

7. Secondary Outcome: (Part 2) Incidence of Adverse Event (AE)s
Description: Number of patients experiencing adverse event (AE)s
Time Frame: throughout study completion, approximately 1 year
Population: Due to early termination of the study, Part 2 and analysis was not conducted.
Arm/Group | BBT-176
Number analyzed (Participants) | 0

8. Secondary Outcome: (Part 2) BBT-176 Concentrations
Description: Plasma BBT-176 concentrations at steady state
Time Frame: At Cycle 2 Day 1 (each cycle is 21 days)
Population: Due to early termination of the study, Part 2 and analysis was not conducted.
Arm/Group | BBT-176
Number analyzed (Participants) | 0

9. Secondary Outcome: (Part 2) Progression Free Survival (PFS)
Description: PFS will be calculated for each patient as the number of days from the first day of treatment to the date of the first documented disease progression or date of death, whichever occurs first.
Time Frame: throughout study completion, approximately 1 year
Population: Due to early termination of the study, Part 2 and analysis was not conducted.
Arm/Group | BBT-176
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Safety monitoring was performed up to 30 days (± 3 days) after the last administration of study drug or immediately before initiation of any other cancer therapies, an average of 6 months.
Description: Due to early termination of the study, analysis was not conducted.
Groups:
- 20mg QD: BBT-176: 20mg, QD, Orally
- 80mg QD: BBT-176: 80mg, QD, Orally
- 160mg QD: BBT-176: 160mg, QD, Orally
- 320mg QD: BBT-176: 320mg, QD, Orally
- 480mg QD: BBT-176: 480mg, QD, Orally
- 600mg QD: BBT-176: 600mg, QD, Orally
- 160mg BID: BBT-176: 160mg, BID, Orally
- 200mg BID: BBT-176: 200mg, BID, Orally
- 240mg BID: BBT-176: 240mg, BID, Orally
Arm/Group | 20mg QD | 80mg QD | 160mg QD | 320mg QD | 480mg QD | 600mg QD | 160mg BID | 200mg BID | 240mg BID
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/3 | 0/8 | 0/3 | 1/5 | 0/9 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 2/4 | 1/3 | 4/8 | 1/3 | 3/5 | 6/9 | 6/6
Other Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 3/4 | 3/3 | 8/8 | 3/3 | 4/5 | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20mg QD (N=4) | 80mg QD (N=3) | 160mg QD (N=4) | 320mg QD (N=3) | 480mg QD (N=8) | 600mg QD (N=3) | 160mg BID (N=5) | 200mg BID (N=9) | 240mg BID (N=6)
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1
COVID-19 related Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20mg QD (N=4) | 80mg QD (N=3) | 160mg QD (N=4) | 320mg QD (N=3) | 480mg QD (N=8) | 600mg QD (N=3) | 160mg BID (N=5) | 200mg BID (N=9) | 240mg BID (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 4 | 3 | 1 | 4 | 5
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 6 | 3 | 1 | 2 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 4 | 3 | 0 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1
Amylase Increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
COVID-19 infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema eyelids (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 4 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early during Part 1, and Part 2 (Phase 2) was not initiated, resulting in no data available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT04820023/Prot_002.pdf
  • Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT04820023/SAP_003.pdf